CLINICAL TRIAL: NCT00336648
Title: A Phase II Pilot Study of Preoperative Gemcitabine and Bevacizumab-Based Chemoradiation for Patients With Resectable Adenocarcinoma of the Pancreas
Brief Title: Preop Chemoradiation Resectable Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0784
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Neoplasms; Bevacizumab; Gemcitabine; Radiation Therapy; adenocarcinoma of the pancreatic head; adenocarcinoma of the uncinate process
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Avastin + Surgery (Experimental): Gemcitabine plus Avastin-based chemoradiation followed by pancreaticoduodenectomy
  Interventions: Drug: Avastin (Bevacizumab); Drug: Gemcitabine; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Avastin (Bevacizumab) — 10mg/kg by vein (IV) on Days 1, 2, 15 and 29 the adjuvant therapy every two weeks starting approximately 6 weeks after surgery for three months.
  Other Names: Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Gemcitabine — 400 mg/m2 IV once a week on Days 1, 2, 8,15, 22, 29, 36 +/-2 days (Saturdays)
  Other Names: Gemcitabine Hydrochloride; Gemzar
Procedure: Radiation Therapy — Day 3 +/-2 days (Monday) Start Radiation therapy, Mon -Fri x 28 days; 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions)
  Other Names: RT; Radiotherapy

SUMMARY:
Primary Objective:

1. To assess resectability rate in patients undergoing gemcitabine plus Avastin-based chemoradiation followed by pancreaticoduodenectomy for adenocarcinoma of the pancreas.

Secondary Objectives:

1. To assess disease free survival and overall survival
2. To assess margin resection rate (R0 vs. R1) in these patients
3. To assess patterns of failure

DETAILED DESCRIPTION:
Gemcitabine is designed to disrupt the growth of the cancer cells, which causes the cancer cells to start to die.

Avastin is designed to prevent or slow down the growth of tumors by its damaging effects on blood vessel growth in tumors.

Before treatment starts, you will have a complete physical exam. Blood (about 2 tablespoons) will be drawn for tests, and a urine test will be performed. Chest x-rays and computed tomography (CT) scans of the abdomen will be done. Women who are able to have children must have a negative blood (1-2 tablespoons) pregnancy test.

If you are found to be eligible to take part in this study, you will receive gemcitabine once a week, Avastin once every 2 weeks, and radiation 5 times a week. Gemcitabine and Avastin will be given on Saturdays, and the radiation will be given Monday through Friday of each week. You will receive this treatment as an outpatient for 6 weeks.

You will receive gemcitabine through a needle in a vein on Days 1, 8, 15, 22, 29, and 36 (+/- 2 days). You will receive Avastin through a needle in a vein every 2 weeks on Days 1, 15, and 29 (+/- 2 days). On the days you receive both drugs, you will receive Avastin over 30-90 minutes and gemcitabine over 40 minutes.

The first dose of Avastin will be given over about 90 minutes. If you do not have a reaction (such as fever/chills), the next dose will be given over about 60 minutes, and if again no reaction occurs, each dose after that will be given over about 30 minutes. If you experience a reaction to the Avastin infusion, you may be given acetaminophen (such as Tylenol) by mouth and/or diphenhydramine (Benadryl) by vein over 30 minutes before each dose to decrease the risk of further reactions.

Radiation will be given Monday through Friday for 5 1/2 weeks. Each day of treatment, you will lie on a treatment table. The radiation therapist will help position your body so that the radiation goes to the right place. A machine will deliver the radiation. It will take about 15-20 minutes to receive the radiation treatment each day.

If any days of radiation are missed, these days will be made up at the end of your treatment (at the end of 28 days) so that you receive the full amount of radiation.

During the study, you will have physical exams weekly while you are receiving chemoradiation, every other week while you are receiving chemotherapy after surgery, and every 4 months during the follow-up period. You will have blood drawn (1-2 tablespoons each time) for routine tests on a weekly basis while you are receiving chemoradiation, every other week while you are taking Avastin after surgery for 3 months, and every 4 months during the follow-up period. The possible development of side effects will be closely monitored and could require extra blood and/or urine samples. You may also have physical exams, blood and urine tests, x-rays, and scans after completing the chemoradiation part of the study, depending upon what is medically needed for evaluation of ongoing therapy.

The overall effect of treatment will be evaluated at least 8 weeks (+/- 2 days) after the completion of chemoradiation. A chest x-ray and CT scans of the chest, abdomen, and pelvis will then be performed, and blood (about 2 tablespoons) will be drawn for routine tests. Some participants will have surgery to remove part of the pancreas, if needed. The reason to wait at least 8 weeks is to allow a safe period of time to pass after the last dose of Avastin to prevent bleeding during surgery. It may also help decrease the risk of postoperative complications, including bleeding and poor wound healing.

This research study allows participants to receive up to 3 infusions of Avastin during the chemoradiation part of the study. If the treatment is shown to benefit you, your doctor may continue to give additional infusions of Avastin every 2 weeks (+/- 2 days) for 3 months after surgery. After the Avastin treatment, you will have a chest x-ray, abdominal CT scan, and blood (about 2 tablespoons) will be drawn for routine tests every 4 months after surgery for 2 years to check the status of the tumor.

This is an investigational study. The study drugs are commercially available and FDA approved, but their use together with radiation is experimental. Avastin is FDA approved for colon and lung cancers but has not been evaluated by the FDA for pancreatic cancer. Gemcitabine is FDA approved for pancreatic cancer. Avastin will be provided free of charge during the study, however the cost of the infusion of the drug will be the responsibility of you and/or your insurance company. The costs of gemcitabine and radiation are considered standard of care, and will be the responsibility of you and/or your insurance company. Up to 31 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreatic head or uncinate process is required prior to treatment. Islet cell tumors are not eligible.
2. Patients must be staged with a physical exam, CXR, and contrast-enhanced CT. Only potentially resectable patients are eligible. Potentially resectable defined as: a) no extra pancreatic disease, b) no evidence (on CT) of tumor extension to the celiac axis or SMA, and c) no evidence (CT or angiogram) of occlusion of the SMV or SMPV confluence. Visceral angiography is optional. Laparoscopic staging is not part of the pretreatment evaluation for this study. Laparoscopy may be performed prior to planned laparotomy at surgeon's discretion. Staging needs to be done within 28 days of enrollment.
3. Patients cannot have known hepatic or peritoneal metastases detected by ultrasound (US), CT scan, or laparotomy prior to chemoradiation.
4. There will be no upper age restriction; patients with Karnofsky performance status greater than 70 are eligible.
5. Adequate renal, and bone marrow function: Leukocytes greater than or equal to 3,000/uL; Absolute neutrophil count greater than or equal to 1,500/uL; Platelets greater than or equal to 100,000/U1; Serum creatinine less than or equal to 2.0-mg/dL and urine protein: creatinine ratio less than or equal to 1.0 at screening
6. Hepatic function (endoscopic or percutaneous drainage as needed) Total bilirubin less than or equal to 2 X institutional upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) less than or equal to 5 X institutional ULN
7. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude protocol therapy.
8. Pregnant women with a positive (blood B-HCG) pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast feeding, as specified in the informed consent.
9. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Tumors in the body or tail of the pancreas (to the left of the portal -SMV confluence) are not eligible.
2. Patients with uncontrolled hypertension, baseline blood pressure of greater than 150/100 mmHg
3. Unstable angina or New York Heart Association (NYHA) Grade II or greater congestive heart failure.
4. History of myocardial infarction, stroke, DVT, or pulmonary embolism within 6 months of the study
5. Clinically significant peripheral vascular disease.
6. Known history of bleeding diathesis coagulopathy. If patient has prior documented PT, INR then INR should be less than 2.0 (patients on anticoagulation for atrial fibrillation, other cardiac disorders, and for remote history of thrombosis are not excluded). Lab results should be within 2 weeks of patient enrollment.
7. Known presence of central nervous system or brain metastases.
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
9. Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
10. Urine protein: creatinine ratio greater than 1.0 at screening; a 24 hour urine protein should be obtained and the level must be less than 1gm/24 hours in order for the patient to be eligible.
11. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
12. Serious, non-healing wound, ulcer, or bone fracture
13. Evidence of duodenal invasion
14. Inability to comply with study and/or follow-up procedures
15. Patients less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Resection | 8 weeks (+/- 2 days) after the completion of chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Evans, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org